CLINICAL TRIAL: NCT04011202
Title: Virtual Reality, Mood, and Sedentary Behaviour After Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19; lack of recruitment; staff turnover.
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Brodie Sakakibara, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VR Stroke
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Stroke; Stroke, Ischemic; Stroke Hemorrhagic; Stroke, Lacunar
Keywords: Stroke; Virtual reality; Depressive symptoms; Sedentary behaviour
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Stroke, Lacunar; Depression

STUDY DESIGN:
Intervention Model Description: Control group and experimental group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Group (Experimental): Receives the VR protocol
  Interventions: Behavioral: Virtual reality gaming program (VR-gaming program)
- Control Group (No Intervention): Receives regular care

INTERVENTIONS:
Behavioral: Virtual reality gaming program (VR-gaming program) — Participants in the VR-gaming program will receive three 20-30 minutes sessions of VR-gaming per week for the duration of their inpatient stay. Participants will select VR games/program in categories of: Relaxation; Leisure sport and activities; or Action/adventure. The VR-gaming program will be implemented one-on-one, face-to-face by a clinician using the commercially-available Oculus Go system.
  Arms: VR Group

SUMMARY:
The purpose of this study is to: 1) evaluate the feasibility (e.g. recruitment and retention, administrative and participant burden) of a VR program to improve mood and sedentary behaviour in inpatient stroke survivors; and 2) develop an understanding of the effects of VR on mood and sedentary behaviours among inpatient stroke survivors.

DETAILED DESCRIPTION:
It is common for individuals who have had a stroke to have deficits in motor and sensory function, communication, and cognition. These deficits pose serious barriers for stroke survivors to effectively manage their health and well-being over time, and has contributed to excessive amounts of sedentary time beginning in inpatient rehabilitation, and continuing post-discharge.

Sedentary behaviours are associated with various health risks. Lying down, sitting for prolonged periods of time, or any other activity with an energy expenditure of ≤1.5 metabolic equivalent units are associated with an increased incident of chronic diseases, as well as with reduced physical function, and increased symptoms of depression and frailty. Moreover, sedentary behaviours are associated with all-cause mortality, with each additional hour spent sedentary increasing mortality risk. Thus, efforts to reduce sedentary time as inpatients may be a promising therapeutic intervention to improve longer term health outcomes of stroke survivors.

Issues with mood after stroke are common. After stroke, depression and depressive symptoms are common occurrences with as many as 28% experiencing depressive disorders or symptoms one month post-stroke, and 36% between two and five months. Similarly, anxiety symptoms and psychological stress are prevalent issues, with 23% reporting anxiety within five months post stroke, and 25% experiencing psychological stress. Not only are these issues associated with reduced quality of life, poorer functional outcomes after rehabilitation, increased healthcare use, and mortality, these psychological factors have also been shown to be associated with sedentary behaviour. It is therefore plausible that decreases in sedentary behaviours may be achieved via mood improvements.

Virtual reality (VR) has garnered substantial attention as a cost-effective treatment approach in stroke rehabilitation, particularly as a means to supplement existing therapy. While the use of VR in stroke rehabilitation has resulted in positive outcomes, the outcomes studied have primarily focused on physical and functional rehabilitation. Despite evidence that VR is emerging as a method to address issues with mood, the use of VR to improve mood among inpatient stroke survivors has yet to be studied.

Objectives: In this research, the investigators will: 1) evaluate the feasibility (e.g. recruitment and retention, administrative and participant burden) of a VR program to improve mood and sedentary behaviour in inpatient stroke survivors; and 2) develop an understanding of the effects of VR on mood and sedentary behaviours among inpatient stroke survivors.

Hypotheses: The investigators expect the protocol will demonstrate sufficient feasibility to support a subsequent larger randomized controlled trial (RCT). The investigators also hypothesize that the VR program will improve the primary endpoints, measures of mood, in people with stroke receiving inpatient rehabilitation, and that such improvements will reduce sedentary behaviour.

This 1-year feasibility study will use a parallel group, single-blinded (tester), randomized controlled trial that will be registered and adhere to the CONSORT guidelines. Eligible participants will be randomly assigned (1:1) to either: 1) Intervention: 3 times per week to discharge of VR-gaming; or 2) Control: usual care.

ELIGIBILITY:
Inclusion Criteria:

* Have had a stroke (confirmed by CT scan or MRI); are an inpatient receiving stroke rehabilitation for an expected length of stay of 14 days or longer; are at least 19 years of age or older; are able to provide informed consent; have clearance from a physician to participate in the study; are able to understand English.

Exclusion Criteria:

* Have a visual or hearing impairment; have a planned surgical intervention; are not medically stable; have a significant musculoskeletal or other neurological condition; severe aphasia.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | Rehabilitation discharge (generally 4-6 weeks)
  The 7-item Depression scale in the Hospital Anxiety and Depression Scale; total sub scale scores range from 0 to 21; higher values indicate more depressive symptoms

SECONDARY OUTCOMES:
Anxiety symptoms | Rehabilitation discharge (generally 4-6 weeks)
  The 7-item Anxiety scale in the Hospital Anxiety and Depression Scale; total sub scale scores range from 0 to 21; higher values indicate more anxiety symptoms
Stress | Rehabilitation discharge (generally 4-6 weeks)
  10-item Perceived Stress Scale; total scores range from 0 to 40; higher values indicate higher perceived stress
Motivation | Rehabilitation discharge (generally 4-6 weeks)
  16-item Situational Motivation Scale, including 4 sub scales: 4-item Instrinsic motivation; 4-item Identified regulation; 4-item External motivation; 4-item Amotivation; Mean sub scale scores are derived, ranging from 1 to 7; higher values indicate higher motivation for each sub scale
Happiness | Rehabilitation discharge (generally 4-6 weeks)
  4-item Subjective Happiness Scale; Mean scores range from 1 to 7; higher values indicate higher happiness
Stroke severity (functional disability) | Rehabilitation discharge (generally 4-6 weeks)
  6-category Modified Ranking Scale; individuals are categorized into one of six categories, ranging from 'no disability = 0' to 'severe disability = 5'. A higher category ranking is indicative of greater disability
Sedentary time | Rehabilitation discharge (generally 4-6 weeks)
  7-item Measure of Older Adults' Sedentary Time; for each item (i.e., sedentary behaviour (e.g., watching tv)), participants estimate the amount of time in that activity in hours and minutes for the past week; total time is summed for an estimated sedentary behaviour for the past week

OTHER OUTCOMES:
Feasibility indicator - recruitment rate | Rehabilitation discharge (generally 4-6 weeks)
  Number of participants recruited per week
Feasibility indicator - retention rate | Rehabilitation discharge (generally 4-6 weeks)
  Number of participants that complete the study, relative to the number that started the study
Feasibility indicator - perceived benefit of the VR Training Program, | Rehabilitation discharge (generally 4-6 weeks)
  17-item study specific Satisfaction survey; Mean scores range from 1 to 5; Higher scores indicate greater satisfaction
Feasibility indicators - treatment fidelity | Rehabilitation discharge (generally 4-6 weeks)
  Percentage of participants that participate in ALL VR Training sessions
Feasibility indicators - participant and tester burden | Rehabilitation discharge (generally 4-6 weeks)
  Percentage of participants that complete a data collection session in 60 minutes or less
Feasibility indicators - trainer burden | Rehabilitation discharge (generally 4-6 weeks)
  Time spent administering each VR session
Feasibility indicators - ease of using equipment | Rehabilitation discharge (generally 4-6 weeks)
  Downtime due to technical difficulties
Feasibility indicators - safety | Rehabilitation discharge (generally 4-6 weeks)
  Number of adverse events due to the VR Training program

CONTACTS AND LOCATIONS:
Overall Officials: Brodie Sakakibara, Principal Investigator — University of British Columbia
Locations (1):
- Kelowna General Hospital, Kelowna, British Columbia, Canada

REFERENCES:
- [Derived] Rash I, Helgason M, Jansons D, Mitchell L, Sakakibara BM. The influence of a virtual reality entertainment program on depressive symptoms and sedentary behaviour in inpatient stroke survivors: a research protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2022 Oct 22;8(1):230. doi: 10.1186/s40814-022-01189-8. PMID 36273223